CLINICAL TRIAL: NCT05717543
Title: Imaging of Corneal and Crystalline by Near Infrared Retro-illumination
Acronym: RETRO-ILLUMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21CH117; 2021-A01496-35 (Other: ANSM)
Record Dates: First submitted 2023-01-26; First posted 2023-02-08 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Eye Diseases
Keywords: pigmentary glaucoma; crystalline pathology; corneal pathology; Retroillumination; Infrared
MeSH Terms: conditions — Eye Diseases; Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: Exploratory pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with corneal pathology, crystalline pathology, or pigmentary glaucoma (Experimental): Patient with corneal pathology, crystalline pathology, or pigmentary glaucoma will be included.
  Imaging by retroillumination will be realized. In case of bilateral disease, both eyes will be photographed
  Interventions: Device: Retro-illuminator

INTERVENTIONS:
Device: Retro-illuminator — The device Retro-illuminator will be used to photograph the eyes.

SUMMARY:
Retroillumination photography is difficult. The reflections on the cornea and the lens are constant and prevent from obtaining a complete and clear image. Study team have modified a slit lamp intended to photograph the anterior segment of the eye in retroillumination by using a light source in the near infrared (780 nm), and a process which eliminates the reflections.

ELIGIBILITY:
Inclusion Criteria:

* Patient with corneal pathology, crystalline pathology, or pigmentary glaucoma with transilluminable iris. In case of bilateral disease, both eyes will be photographed
* Patient having received an instillation of eye drops to dilate the pupil of the eye to be photographed (or of both eyes).

Exclusion Criteria:

* Major blepharospasm
* Poor or no pupillary dilation: patient with allergy or intolerance to eye drops used for pupillary dilation, refusal of pupillary dilation
* Pregnant or breastfeeding patient
* Person under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Percentage of pictures without reflection (%) | Year: 1
  Evaluation of the device's retroillumination. Pictures without reflection: no reflection or a minimal reflection without loss of information.

SECONDARY OUTCOMES:
Percentage of pictures clean on the pathological area (%) | Year: 1
  Evaluation of the device's retroillumination. Pictures clean : absence of blur, or minimal blurred that does not result in loss of information..
Serious adverse events | Year: 1
  Number of serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Gilles THURET, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No